CLINICAL TRIAL: NCT05674851
Title: Study and Modeling of Organ Motion During Abdominal Imaging
Brief Title: Modeling Organ Motion During Abdominal Imaging in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00111970
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteers
Keywords: Magnetic Resonance Imaging (MRI); Abdominal Cancer; Radiation Therapy Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteer MRI (Experimental)
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — collection of MRI scans for mathematical model development

SUMMARY:
In this study, we plan to systematically analyze the motion of organs and tissues in the abdomen, to understand the physical mechanisms of three-dimensional (3D) motion and interactions of abdominal organs and tissues. This work will allow us to learn how to mathematically model and predict abdominal organ motion.

DETAILED DESCRIPTION:
Specifically, we plan to conduct this study in 3 steps, in an order of increasing complexity, starting with the (intra-fractional) respiratory only motion, then adding intra-fractional GI motility motion, and finally the inter-fractional anatomical variations (adding food intakes and fecal excretion). The research methods described will allow the study team to develop the ability to estimate the motion of both tumor target and critical organs given the patient's MRI, CBCT or x-ray fluoroscopy images on the day of radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* No contraindications for MRI (e.g., unsafe MRI implanted devices, shrapnel, history of metal fragments in eyes, neurostimulators, body habitus, claustrophobia).
* May have pre-existing medical conditions provided they are capable of completing the exam and their condition is not expected to affect the physical tissue properties of the organs that will be imaged.
* Women of child-bearing potential must verbally confirm lack of pregnancy prior to signing consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
abdominal respiratory motion as measured by MRI | baseline
gastrointestinal motility motion as measured by MRI | baseline
inter-fractional motion as measured by MRI | baseline, up to 6 months
  inter-fractional motion is defined as the change in motion of organs and tissues between different image examinations on different days

CONTACTS AND LOCATIONS:
Overall Officials: John Ginn, PhD, Principal Investigator — Duke University Health System (DUHS); Deshan Yang, PhD, Principal Investigator — Duke University Health System (DUHS)
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No